CLINICAL TRIAL: NCT06868836
Title: A Phase II Study of JS207 (PD-1/VEGF Bispecific Antibody) in Combination With Pemetrexed and Platinum in Advanced Non-small Cell Lung Cancer With Actionable Genomic Alterations and TKI Therapy Failure
Brief Title: A Study of JS207 (PD-1/VEGF Bispecific Antibody) in Combination With Chemotherapy in Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS207-002-II-NSCLC
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: JS207 (10 mg/kg or 15 mg/kg, IV, d1) + pemetrexed (500 mg/m², IV, d1) + platinum-based chemotherapy (carboplatin: AUC5, d1 or cisplatin 75 mg/m², d1) every 3 weeks (Q3W) for a total of 4 cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS207 + pemetrexed+ platinum-based chemotherapy (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: JS207; Drug: Pemetrexed; Drug: Carboplatin or cisplatin

INTERVENTIONS:
Drug: JS207 — JS207 (10 mg/kg or 15 mg/kg, IV, d1)
Drug: Pemetrexed — Pemetrexed (500 mg/m², IV, d1)
Drug: Carboplatin or cisplatin — Platinum-based chemotherapy (carboplatin: AUC5, d1 or cisplatin 75 mg/m², d1) every 3 weeks (Q3W) for a total of 4 cycles

SUMMARY:
This study targets patients with advanced NSCLC driven with positive driver genes who have failed TKI treatment, enrolling 36-42 participants. Patients will receive JS207 (10 or 15 mg/kg, IV, d1) + pemetrexed (500 mg/m², IV, d1) + platinum-based chemotherapy (carboplatin AUC5 or cisplatin 75 mg/m², d1) every 3 weeks for 4 cycles. Afterward, JS207 and pemetrexed will continue as maintenance therapy until discontinuation criteria are met. The study aims to assess the safety, tolerability, and preliminary efficacy of JS207 combination therapy.

DETAILED DESCRIPTION:
This study enrolls patients with advanced non-small cell lung cancer (NSCLC) who have positive driver genes and have failed TKI treatment. Approximately 36-42 patients are expected to be enrolled and receive treatment with JS207 (10 mg/kg or 15 mg/kg, IV, d1) + pemetrexed (500 mg/m², IV, d1) + platinum-based chemotherapy (carboplatin: AUC5, d1 or cisplatin 75 mg/m², d1) every 3 weeks (Q3W) for a total of 4 cycles.After the 4 cycles, patients will continue receiving JS207 (10 mg/kg or 15 mg/kg, IV, d1) + pemetrexed (500 mg/m², IV, d1) every 3 weeks (Q3W) until they meet the criteria for treatment discontinuation.The study aims to evaluate the safety, tolerability, and preliminary efficacy of JS207 in combination with pemetrexed and platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old (both 18 and 75 years old included) at the time of signing the informed consent form, applicable to both males and females.
2. Locally advanced (stage IIIB/IIIC), metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC) confirmed by histology or cytology, which is not eligible for radical surgery or radical chemoradiotherapy.
3. Positive for driver gene and having received the first-line targeted therapy approved by the National Medical Products Administration (NMPA).
4. Failure of previous tyrosine kinase inhibitor (TKI) treatment and currently having no standard TKI treatment available.
5. Positive for PD-L1 (tumor proportion score, TPS ≥ 1%) confirmed by the central laboratory test or local test.
6. Being able to provide a qualified test report for positive driver gene, or agreeing to provide a qualified sample for driver gene testing.
7. According to the RECIST v1.1 criteria, the subject has at least 1 measurable lesion.
8. Performance status score of 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
9. Expected survival period ≥ 12 weeks.
10. The function of important organs meets the requirements of the protocol.
11. Female subjects of childbearing potential, and male subjects whose partners are females of childbearing age, need to adopt a highly effective contraceptive measure during the study treatment period and for at least 6 months after the last administration.
12. Voluntarily joining this study, signing the informed consent form, having good compliance, and cooperating with the follow-up.

Exclusion Criteria:

1. Diseases accompanied by those listed in the protocol, including those with histopathological or cytopathological confirmation of the tumor combined with neuroendocrine tumor (including small cell lung cancer, large cell neuroendocrine carcinoma, etc.) components, or with the squamous cell carcinoma component exceeding 10%; known meningeal metastasis; symptomatic brain metastasis; the tumor encircling important blood vessels or with obvious necrosis and cavities, and the investigator deems that it may pose a risk of bleeding, etc.
2. Treatment received as listed in the protocol, including immunologically mediated treatment; drugs targeting the anti-VEGF pathway, etc.
3. Having an obvious bleeding tendency or a history of severe coagulation dysfunction.
4. Gastrointestinal perforation, intra-abdominal fistula or intra-abdominal abscess occurred within 6 months before the first administration, or currently having high-risk factors for perforation/fistula formation of the hollow viscus as judged by the investigator.
5. Having a serious, unhealed or ruptured wound, active ulcer or untreated fracture.
6. Having uncontrolled hypertension, or a history of hypertensive crisis or hypertensive encephalopathy.
7. Expected that the toxicity of previous anti-tumor treatment has not recovered to ≤ grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE).
8. Known allergy to the investigational drug or its excipients, pemetrexed, platinum drugs (carboplatin/cisplatin), or known history of ≥ grade 3 allergy to antibody drugs in the past.
9. Having an active autoimmune disease or a history of autoimmune disease.
10. Having a history of immunodeficiency.
11. Having a severe infection within 4 weeks before the first use of the investigational drug.
12. History of confirmed or suspected interstitial lung disease, idiopathic pulmonary fibrosis, drug-induced pneumonia, idiopathic pneumonia, or other moderate to severe lung diseases that seriously affect lung function.
13. Active pulmonary tuberculosis infection detected by medical history or CT examination.
14. Having active tuberculosis, hepatitis B, or hepatitis C.
15. Having been diagnosed with any other malignant tumor within 5 years before the first use of the investigational drug.
16. Uncontrolled concurrent diseases listed in the protocol.
17. As judged by the investigator, having other severe, acute or chronic medical diseases, mental diseases or laboratory abnormalities that may increase the risk associated with participating in the study, or may interfere with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed objective response rate (ORR) | Up to approximately 25 months
  Evaluate the investigator-assessed objective response rate (ORR) of JS207 combined with pemetrexed and platinum-based chemotherapy in the treatment of advanced non-squamous non-small cell lung cancer (NSCLC) patients with positive driver genes and who have failed tyrosine kinase inhibitor (TKI) therapy.The ORR is defined as the proportion of subjects who have a partial response (PR) or a complete response (CR) in the Best Overall Response

SECONDARY OUTCOMES:
Investigator-assessed objective response rate (DCR) | Up to approximately 25 months
  The DCR is defined as the proportion of subjects whose Best Overall Response (BOR) is Complete Response (CR), Partial Response (PR), or Stable Disease (SD)
Investigator-assessed Duration of Response (DoR) | Up to approximately 25 months
  The DoR is defined as the time from the first occurrence of CR or PR to the first occurrence of Progressive Disease (PD) or death (whichever occurs first). The DoR is only applicable to subjects whose BOR is CR or PR
Investigator-assessed Progression-Free Survival (PFS) | Up to approximately 25months
  The PFS is defined as the time from the first administration of the drug to the first documented disease progression (PD) according to the RECIST v1.1 criteria or death due to any disease (whichever occurs first)
Investigator-assessed overall survival (OS) | Up to approximately 25 months
  The OS is defined as the time from the first administration of the drug to death due to any cause
Adverse Event | Up to approximately 25 months
  Collect Serious Adverse Events (SAEs) and Adverse Events (AEs) from the time of signing the Informed Consent Form (ICF) until the safety follow-up visit.Evaluate the safety of the investigational drug
Number of participants with Laboratory examination indices | Up to approximately 25 months
  Collect all laboratory examinations during the study period or the safety follow-up period. The investigator must review the laboratory examination results, record the review findings, and record any clinically significant changes that occur during the study period as Adverse Events. Evaluate the safety of the investigational drug

OTHER OUTCOMES:
the trough concentrations (PK) | Up to approximately 25 months
  To characterize the trough concentrations of JS207
Immunogenicity(ADA) | Up to approximately 25 months
  The immunogenicity of JS207, including the titer of ADA
Immunogenicity(NAb) | Up to approximately 25 months
  The immunogenicity of JS207, including the incidence rate of neutralizing antibodies (NAb) (if applicable)
Expression level of PD-L1 in tumor tissues | Up to approximately 5 months
  The correlation between the expression level of PD-L1 in tumor tissues and the therapeutic effect

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Wang, Doctor, Study Director — Medical Director
Locations (1):
- Guangdong Provicial People's Hospital, Guangzhou, Guangdong, China